CLINICAL TRIAL: NCT01404637
Title: The Effects of Tamsulosin 0.4mg on Clinical Outcomes in Korean Men With Severe Symptomatic BPH
Brief Title: Effects of Tamsulosin 0.4mg on Clinical Outcomes in Korean Men With Severe Symptomatic Benign Prostatic Hyperplasia (BPH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sung Won Lee MD, Ph.D, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-02-052
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Tamsulosin 0.4mg (Experimental)
  Interventions: Drug: Tamsulosin 0.4mg
- tamsulosin 0.2mg (Active Comparator)
  Interventions: Drug: Tamsulosin 0.2mg

INTERVENTIONS:
Drug: Tamsulosin 0.4mg — Treatment: tamsulosin 0.2mg (2T) /day Posology: two 0.2 mg tablet to be taken after an evening meal.
  Arms: Tamsulosin 0.4mg
Drug: Tamsulosin 0.2mg — tamsulosin 0.2mg (1T) /day Posology: one tablet to be taken after an evening meal.
  Arms: tamsulosin 0.2mg

SUMMARY:
The purpose of this study is to compare the efficacy and safety of tamsulosin 0.4mg (Harnal® D. 0.2mg, 2T) with tamsulosin 0.2mg (Harnal® D 0.2mg, 1T) in patients with severe symptomatic benign prostatic hyperplasia as a first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe LUTS : IPSS ≥ 20

Exclusion Criteria:

* Post voided residual urine ≥ 150mL
* Patients performing catheterization
* Urinary tract infection patients
* Patients taking 5 alpha reductase inhibitor
* Known hypersensitivity to tamsulosin
* History of postural hypotension or syncope
* Hypertension patients treated with other alpha1-blockers
* Patients newly taking anticholinergic medication within 1 month
* Hepatic insufficiency (AST/ALT ≥ 2 times of normal range)
* Renal insufficiency (s-Cr ≥ 2mg/dL)

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Changes of the total International Prostate Symptom Score (IPSS) score from baseline to 12 weeks of treatment in patients with severe symptomatic BPH refractory to tamsulosin 0.2mg (Harnal® 0.2mg, 1T) | 12 weeks of treatment

SECONDARY OUTCOMES:
Changes of maximal flow rate and post-voided residual urine volume after 4 and 12 weeks treatment. | 4 weeks and 12 weeks of treatment
Changes of parameters in voiding diary after 4 and 12 weeks treatment. | 4 weeks and 12 weeks of treatment

REFERENCES:
- [Derived] Kim JJ, Han DH, Sung HH, Choo SH, Lee SW. Efficacy and tolerability of tamsulosin 0.4 mg in Asian patients with lower urinary tract symptoms secondary to benign prostatic hyperplasia refractory to tamsulosin 0.2 mg: a randomized placebo controlled trial. Int J Urol. 2014 Jul;21(7):677-82. doi: 10.1111/iju.12412. Epub 2014 Apr 13. PMID 24725169